CLINICAL TRIAL: NCT03669627
Title: A Randomized Controlled Observer Blind Trial to Compare the Immunogenicity and Acceptability of a MF59-adjuvanted Influenza Vaccine Compared to an Inactivated Influenza Vaccine as a Preferred Influenza Vaccine Priming Strategy for Naive Infants 6 to <24 Months of Age
Brief Title: CT18 Infant Influenza Priming Study in Vaccine Naive Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Immunization Research Network (Network)
Collaborators: Provincial Health Services Authority British Columbia (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Université de Montréal (Other); Canadian Center for Vaccinology (Other); CHU de Quebec-Universite Laval (Other); Dalhousie University (Other)
Responsible Party: Principal Investigator, Joanne Langley, Principal Investigator, Canadian Immunization Research Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CT18
Record Dates: First submitted 2018-09-05; First posted 2018-09-13 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Influenza
Keywords: infants; priming; Fluad; Fluzone
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three groups: Group 1 will receive aTIV as a primer and QIV as a booster, Group 2 will receive QIV as both primer and booster, and Group 3 will receive aTIV as both primer and booster.
Who Masked: Investigator
Masking Description: Observer-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: aTIV primer, QIV booster (Active Comparator): Two doses (0.25 mL) aTIV (FLUAD )received one month apart in year 1. One dose (0.5 mL) QIV (Fluzone) received as booster in year 2.
  Interventions: Biological: aTIV Primer; Biological: QIV Booster
- Group 2: QIV primer, QIV booster (Other): Standard of care control group:
  Two doses (0.5 mL) QIV (Fluzone) received one month apart in year 1. One dose (0.5 mL) QIV (Fluzone) received as booster in year 2.
  Interventions: Biological: QIV Primer; Biological: QIV Booster
- Group 3: aTIV primer, aTIV booster (Experimental): This arm is experimental in that some participants will be receiving the MF59-adjuvanted TIV (FLUAD) in year two of the study, after the age of two years, which is off label.
  Two doses (0.25 mL) TIV (FLUAD) received one month apart in year 1. One dose (0.25 mL) TIV (FLUAD) received as booster in year 2.
  Interventions: Biological: aTIV Primer; Biological: aTIV Booster

INTERVENTIONS:
Biological: aTIV Primer — MF59-adjuvanted trivalent influenza virus primer: 2 doses (0.25mL) one month apart
  Other Names: FLUAD Pediatric®
  Arms: Group 1: aTIV primer, QIV booster; Group 3: aTIV primer, aTIV booster
Biological: QIV Primer — Unadjuvanted quadrivalent influenza vaccine primer: 2 doses (0.5mL) one month apart
  Other Names: Fluzone® Quadrivalent
  Arms: Group 2: QIV primer, QIV booster
Biological: aTIV Booster — MF59-adjuvanted influenza virus vaccine booster: 1 dose (0.25mL), year 2
  Other Names: FLUAD Pediatric®
  Arms: Group 3: aTIV primer, aTIV booster
Biological: QIV Booster — Unadjuvanted quadrivalent influenza vaccine booster: 1 dose (0.5mL), year 2
  Other Names: Fluzone® Quadrivalent
  Arms: Group 1: aTIV primer, QIV booster; Group 2: QIV primer, QIV booster

SUMMARY:
This study evaluates whether priming influenza naive infants, age six to 23 months, with a MF59-adjuvanted (oil in water emulsion) influenza vaccine is preferred to priming with an inactivated unadjuvanted influenza vaccine. All participants will receive a priming vaccine, either MF59-adjuvanted trivalent influenza vaccine (aTIV) or unadjuvanted quadrivalent influenza vaccine (QIV). For the booster shot the following year, two thirds of participants will receive QIV and one third will receive MF59-adjuvanted vaccine.

DETAILED DESCRIPTION:
Children under 24 months of age suffer from an influenza burden (high morbidity and mortality) similar to that of the elderly, and have been identified as a high priority target for vaccination programs by Canada's National Advisory Committee on Immunization. There is evidence that a person's first exposure to influenza antigens may have long-term implications for protection.

This is a randomized, controlled, observer-blind study that will assign participants to one of three groups. Group 1 will receive MF59-adjuvanted influenza vaccine (two doses one month apart) in the fall of year 1, followed by QIV (one dose) in the fall of year 2. Group 2 will receive QIV (two doses one month apart) in the fall of year 1, followed by QIV (one dose) in the fall of year 2. Group 3 will receive MF59-adjuvanted IV (two doses one month apart) in the fall of year 1, followed by MF59-adjuvanted IV (one dose) in the fall of year 2.

ELIGIBILITY:
Inclusion Criteria:

* Parent/LAR is willing and able to give informed consent for participation in the trial.
* Male or Female, aged six months to 23 months.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.

Exclusion Criteria:

* Any significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participant in another research trial involving an investigational product or medical device in the prior 12 weeks.
* Prior receipt of an influenza vaccine
* History of laboratory-confirmed influenza infection, by parent/LAR report
* Hypersensitivity to any vaccine component of products used in this study (see product monographs)
* Immunodeficiency or autoimmune disease

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Serum hemagglutination inhibition (HI) antibody titers | Before and after priming with the various vaccine combinations at day 393.
  Serum HI antibodies to influenza antigens A/H3N2, A/H1N1, and B Yamagata and Victoria lineages will be used to calculate the seroconversion rate and the seroprotection rates.

SECONDARY OUTCOMES:
Adverse Events (AEs) | Days 0 to 545
  Measure local and systemic solicited and unsolicited adverse events following each vaccine dose, and severe AE throughout the study.

OTHER OUTCOMES:
Vaccine acceptability: parent/Legally Authorized Representative (LAR) questionnaire | Days 56, 180, 393, and 545
  The Acceptability Questionnaire measures parental opinions about side effects of the study vaccines. There are four questions with a scale range evaluating degree of certainty and one open-ended question with a free text response. There is no total score.
Cell-Mediated Immunity | Days 0, 56, 180, 365, 393, 545
  To assess cell mediated immune responses to three influenza immunization two priming schedules in vaccine naïve infants.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Langley, MD, Principal Investigator — Dalhousie University, Canadian Center for Vaccinology; Soren Gantt, MD, PhD, Principal Investigator — BC Children's Hospital, UBC
Locations (4):
- Canada (4):
  - Vaccine Evaluation Center, BC Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - Research Institute of the McGill University health Centre, Montreal, Quebec
  - Équipe de recherche en vaccination CHU de Québec-Université Laval, Québec, Quebec